CLINICAL TRIAL: NCT01253720
Title: PACE CALL: A Tailored Weight Management Program for Childhood ALL Survivors
Brief Title: PACE CALL: Weight Loss Study for Childhood Leukemia Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huang, Jeannie, M.D. (Individual)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 070731
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-03

CONDITIONS: Acute Lymphoblastic Leukemia; Cancer; Obesity
Keywords: obesity; text messages; internet; cancer; overweight
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms; Obesity; Overweight

ARMS (2):
- PACE CALL/Fit4Life (Experimental): Fit4Life intervention activities:
  Website: Provides weekly nutrition, physical activity, and weight loss information.
  Counseling Calls: Participants and their parents will get phone calls from their Health Coach to assess progress & problems.
  Health Coach Question & Answer: Participants will be assigned a Health Coach that they can contact at any time to ask questions or express any concerns.
  Text & Picture Messages: Participants will receive daily text messages to help remind them of being healthy. Messages will relate to the weekly topics and general checking in questions.
  Parent Materials: Parents will receive a packet of printed materials that relate to parenting skills regarding being a healthy role model for their child and healthy eating and exercise tips.
  Interventions: Behavioral: PACE CALL/Fit4Life
- Control (No Intervention): The Control group will receive monthly mailings on basic nutrition and physical activity information.

INTERVENTIONS:
Behavioral: PACE CALL/Fit4Life — The Fit4Life E intervention will be designed to promote weight loss and subsequent weight loss maintenance through the adoption and maintenance of improved eating, physical activity and sedentary behaviors in at risk for overweight and overweight adolescent survivors of ALL and their parent/guardian. the Fit4Life intervention will incorporate elements of the Chronic Care Model, including frequent phone and mail interactions, an initial in-person encounter to provide encouragement and initial patient-tailored counseling for obesity management, family-centered skill development to achieve healthy behavioral modification via goal setting, self-monitoring, and problem solving.
  The Fit4Life intervention includes:
  Web-based weight loss program Text and Picture messages Counseling Calls Health Coach
  Arms: PACE CALL/Fit4Life

SUMMARY:
UC San Diego researchers conducted a study to develop and evaluate an internet and text message based weight loss study for childhood acute lymphoblastic leukemia (ALL) survivors. We hypothesized that those study participants randomized to the intervention will demonstrate greater reduction in BMI-z score as compared to the control group.

DETAILED DESCRIPTION:
The PACE CALL or Fit4Life study, sponsored by the American Cancer Society , was a 4-year research project aimed at developing and testing the efficacy of a web & cell phone based weight loss program. The purpose of the intervention was to promote weight loss and management and improve physical activity, diet and sedentary behaviors among preadolescent and adolescent youth (7-18) who are survivors of childhood ALL (defined as being off therapy for at least 2 years without disease relapse). Fit4Life was based on and adapted from notable prior successful adolescent weight control interventions, and physical activity and diet behavioral promotion interventions in the preadolescent and adolescent age group. Particular sensitivity to issues experienced by cancer survivors and their families were incorporated into this newly developed intervention based on systematic cancer survivor input and feedback as well as mentor/collaborator input regarding cancer survivor research.

ELIGIBILITY:
Inclusion Criteria:

* 7 - 18 years old
* survived childhood acute lymphoblastic leukemia (defined as being off treatment for at least 2 years)
* greater than or equal to 85th percentile BMI-for-age and gender)
* read and speak English
* have a parent that reads and speaks English or Spanish
* willingness to attend assessments
* access to the Internet

Exclusion Criteria:

* any comorbidities of obesity that require immediate sub-specialist referral including pseudotumor cerebri, sleep apnea, and obesity hypoventilation syndrome
* any subject with a known disease of the liver, pancreas or small intestine that would adversely effect digestion or absorption of nutrients
* any pulmonary, cardiovascular, orthopedic, or musculoskeletal problem that would limit ability to adhere to moderate-level physical activity recommendations
* have a history of substance abuse or other psychiatric disorder that would impair compliance with the study protocol
* are using any medications which alter body weight
* are currently enrolled in another weight loss program
* in foster care

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2008-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
BMI | Baseline, 4 months
  To determine the impact of a weight loss intervention on BMI compared to a control group

SECONDARY OUTCOMES:
Weight Loss Behaviors | Baseline, 4 months
  To determine the impact of a weight loss intervention vs. a control group on self-reported behavioral measures of diet and physical activity.
Metabolic Blood Measures | Baseline, 4 months
  To determine the impact of a weight loss intervention vs. control on fasting serum insulin, fasting blood glucose, and blood lipid levels.
Psychosocial Mediators of Weight Loss Behaviors | Baseline, 4 months
  To determine the impact of a weight loss intervention vs. control on psychosocial mediators of diet and physical activity behavior changes
Quality of Life | Baseline, 4 months
  To determine the impace of a weight loss intervention vs. control on quality of life and depression.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

REFERENCES:
- [Result] Huang JS, Dillon L, Terrones L, Schubert L, Roberts W, Finklestein J, Swartz MC, Norman GJ, Patrick K. Fit4Life: a weight loss intervention for children who have survived childhood leukemia. Pediatr Blood Cancer. 2014 May;61(5):894-900. doi: 10.1002/pbc.24937. Epub 2014 Jan 16. PMID 24436138